CLINICAL TRIAL: NCT04796896
Title: A Phase 2/3, Three-Part, Open-Label, Dose-Escalation, Age De-escalation and Randomized, Observer-Blind, Placebo-Controlled Expansion Study to Evaluate the Safety, Tolerability, Reactogenicity, and Effectiveness of mRNA-1273 SARS-CoV-2 Vaccine in Healthy Children 6 Months to Less Than 12 Years of Age
Brief Title: A Study to Evaluate Safety and Effectiveness of mRNA-1273 COVID-19 Vaccine in Healthy Children Between 6 Months of Age and Less Than 12 Years of Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1273-P204
Record Dates: First submitted 2021-03-11; First posted 2021-03-15 (Actual); Results first posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts 1 and 3 are Open-label; Part 2 Randomized and Observer-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mRNA-1273 (Experimental): Part 1: Participants will receive 2 IM injections of mRNA-1273 at doses pre-specified for this study, on Days 1 and 29. Participants will be offered an optional BD of mRNA-1273 lower than the dose chosen for primary series, ≥6 months after Dose 2. After protocol amendment (PA) 9, participants who have not yet received a BD will be offered a BD with mRNA-1273.214.
  Part 2: Participants will receive 2 IM injections of mRNA-1273 at dose selected from Part 1 on Days 1 and 29. Participants (6 to <12 year) will be offered an optional BD of mRNA-1273 lower than the dose chosen for primary series, ≥6 months after Dose 2. After PA 9, participants who have not yet received a BD will be offered a BD with mRNA-1273.214.
  Part 3: Participants will receive 2 IM injections of mRNA-1273 on Days 1 and 29 as primary series then 1 IM injection as Dose 3, on Day 149 ≥3 months and ≤5 months after receipt of Dose 2 of primary series. All 3 injections will be administered at lower dose than that of Part 1.
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.214
- Placebo (Placebo Comparator): Part 2 only: Participants will receive 2 IM injections of mRNA-1273-matching placebo on Day 1 and Day 29. Participants (6 to <12 year old) will be offered an optional BD of mRNA-1273 at a dose lower than the dose that was chosen for the primary series for this age group, at least 6 months post-cross-over Dose 2. After PA 9, participants who have not yet received a BD will be offered a BD with mRNA-1273.214.
  Interventions: Biological: mRNA-1273; Biological: Placebo; Biological: mRNA-1273.214

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo
Biological: mRNA-1273.214 — Sterile liquid for injection

SUMMARY:
The primary goal for this study is to evaluate up to 3 dose levels of mRNA-1273 vaccine given to healthy children as intramuscular (IM) injection in 2 doses (in Parts 1 and 2) and 3 doses (in Part 3), and a third dose or an optional booster dose (BD) (in Parts 1 and 2).

DETAILED DESCRIPTION:
This is a Phase 2/3, 3-part, open-label, dose-escalation, age de-escalation, randomized, observer-blind, placebo-controlled, expansion study intended to infer the effectiveness of mRNA-1273 in children aged 6 months to less than 12 years.

Please access http://www.kidcovestudy.com for additional information, such as Study Overview, Participation, Site Locations along with contact numbers for each location for the study.

ELIGIBILITY:
Key Inclusion Criteria:

* For participants with chronic diseases (such as, asthma, diabetes mellitus, cystic fibrosis, human immunodeficiency virus [HIV] infection), the disease should be stable, per investigator assessment.
* Investigator assessment that the parent(s)/legally acceptable representatives understand and are willing and physically able to comply with protocol mandated follow-up, including all procedures, written informed consent is provided, and participants provide assent.
* For children 2 years of age or older has a body mass index at or above the third percentile according to World Health Organization (WHO) Child Growth Standards at the Screening Visit.
* For children 6 months to <12 months of age: born at full-term with a minimum birth weight of 2.5 kilograms (kg).
* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first injection, agreement to continue adequate contraception or abstinence through 3 months following the second injection (Day 29) and the third dose in Part 3 (Day 149/booster dose Day 1), and not currently breastfeeding.

Key Exclusion Criteria:

* Known history of SARS-CoV-2 infection within 2 weeks prior to administration of vaccine or known close contact with anyone with laboratory-confirmed SARS-CoV-2 infection or COVID-19 within 2 weeks prior to administration of vaccine.
* Prior administration of an investigational or approved CoV (such as, SARS-CoV-2, SARS CoV, Middle East Respiratory Syndrome CoV) vaccine.
* Treatment with investigational or approved agents for prophylaxis against COVID 19 (such as, receipt of SARS-CoV-2 monoclonal antibodies) within 6 months prior to enrollment.
* Known hypersensitivity to a component of the vaccine or its excipients.
* A medical or psychiatric condition that, according to the investigator's judgment, may pose additional risk as a result of participation, interfere with safety assessments, or interfere with interpretation of results.
* History of a diagnosis or condition that, in the judgment of the investigator, may affect study endpoint assessment or compromise participant safety.
* Received any non-study vaccine within 14 days before or after any dose of vaccine (except for seasonal influenza vaccine, which is not permitted within 14 days before or after any dose of vaccine)
* Received intravenous or subcutaneous blood products (red blood cells, platelets, immunoglobulins) within 3 months prior to Day 1
* Participated in an interventional clinical study within 28 days prior to Day 0 or plans to donate blood products while participating in this study.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 11942 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (83):
  - Children's of Alabama, Birmingham, Alabama
  - MedPharmics, LLC, Phoenix, Arizona
  - Emmaus Research Center Inc, Anaheim, California
  - Velocity Clinical Research - Banning - ERN- PPDS, Banning, California
  - SeraCollection Research Services LLC, El Monte, California
  - UCSD Altman Clinical and Translational Research Institute Building, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Rady Childrens Hospital San Diego - PIN, San Diego, California
  - Carey Chronis MD Pediatric, Infant and Adolescent Medicine - FOMAT, Ventura, California
  - Children's Hospital Colorado - (CRS), Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Prohealth Research Center, Doral, Florida
  - University of Florida Jacksonville, Jacksonville, Florida
  - Kissimmee Clinical Research (KCR), Kissimmee, Florida
  - Allied Biomedical Research Institute, Miami, Florida
  - Pensacola Research Consultants Inc. d/b/a Avanza Medical Research Center, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Iresearch Atlanta, LLC, Decatur, Georgia
  - iresearch Savannah, Savannah, Georgia
  - Velocity Clinical Research - Boise - ERN - PPDS, Meridian, Idaho
  - Ann and Robert H Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - Alliance for Multispecialty Research -El Dorado, El Dorado, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Michael W Simon, MD PSC, Lexington, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Pennington Biomedical Research Center, Baton Rouge, Louisiana
  - MedPharmics - Platinum, Metairie, Louisiana
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Javara Inc., Chevy Chase, Maryland
  - The Pediatric Centre of Frederick, Frederick, Maryland
  - Tufts University - Boston - PPDS, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Pediatric Associates of Fall River, Fall River, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - University of Minnesota Masonic Children's Hospital, Minneapolis, Minnesota
  - MediSync Clinical Research Hattiesburg Clinic, Petal, Mississippi
  - University of Missouri Health Care System, Columbia, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Meridian Clinical Research (Hastings, Nebraska), Hastings, Nebraska
  - Meridian Clinical Research (Norfolk-Nebraska) - Platinum - PPDS, Norfolk, Nebraska
  - Quality Clinical Research - PPDS, Omaha, Nebraska
  - MedPharmics, LLC, Albuquerque, New Mexico
  - University of New Mexico, Albuquerque, New Mexico
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Binghamton, New York
  - Certified Research Associates, Cortland, New York
  - Child Healthcare Associates - East Syracuse, East Syracuse, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Javara Inc. - Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center - PIN, Cincinnati, Ohio
  - Lynn Health Science Institute - ERN - PPDS, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Velocity Clinical Research - Providence - ERN - PPDS, Warwick, Rhode Island
  - Coastal Pediatric Associates, Charleston, South Carolina
  - Medical University of South Carolina- PPDS, Charleston, South Carolina
  - Palmetto Pediatrics, North Charleston, South Carolina
  - Meharry Medical College - Clinical and Translational Research Center & Meharry Medical College - Pediatric Department, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Tekton Research - Texas - Platinum - PPDS, Austin, Texas
  - BRCR Global Texas, Edinburg, Texas
  - Pininos Pediatric Services, El Paso, Texas
  - Ventavia Research Group - Platinum - PPDS, Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - West Houston Clinical Research - Hunt, Houston, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Cyfair Clinical Research Center - ERN- PPDS, Houston, Texas
  - Village Health Partners - HUNT, Plano, Texas
  - Victoria Clinical Research, Port Lavaca, Texas
  - Javara, Inc., The Woodlands, Texas
  - Crossroads Clinical Research (Victoria), Victoria, Texas
  - Tanner Clinic, Layton, Utah
  - Advanced Clinical Research/Velocity Clinical Research, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - University of Wisconsin - Madison, Madison, Wisconsin
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Winnipeg Children's Hospital, HSC-Winnipeg, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation - Clinic/Outpatient Facility, Toronto, Ontario
  - McGill University Health Centre-Vaccine Study Centre, Pierrefonds, Quèbec

REFERENCES:
- [Derived] Rostad CA, Campbell JD, Paulsen GC, Ghamloush SS, Xu W, Zheng L, McElrath MJ, De Rosa SC, Girard B, Das R, Anderson EJ, Creech CB. Evaluation of Cellular Immune Responses After mRNA-1273 Vaccination in Children 6 Months to 11 Years of Age. J Infect Dis. 2025 Jun 2;231(5):e945-e955. doi: 10.1093/infdis/jiaf144. PMID 40119775
- [Derived] Berthaud V, Creech CB, Rostad CA, Carr Q, de Leon L, Dietrich M, Gupta A, Javita D, Nachman S, Pinninti S, Rathore M, Rodriguez CA, Luzuriaga K, Towner W, Yeakey A, Brown M, Zhao X, Deng W, Xu W, Zhou H, Girard B, Kelly R, Slobod K, Anderson EJ, Das R, Miller J, Schnyder Ghamloush S. Safety and Immunogenicity of an mRNA-1273 Booster in Children. Clin Infect Dis. 2024 Dec 17;79(6):1524-1532. doi: 10.1093/cid/ciae420. PMID 39158584
- [Derived] Anderson EJ, Creech CB, Berthaud V, Piramzadian A, Johnson KA, Zervos M, Garner F, Griffin C, Palanpurwala K, Turner M, Gerber J, Bennett RL, Ali K, Ampajwala M, Berman G, Nayak J, Chronis C, Rizzardi B, Muller WJ, Smith CA, Fuchs G, Hsia D, Tomassini JE, DeLucia D, Reuter C, Kuter B, Zhao X, Deng W, Zhou H, Ramirez Schrempp D, Hautzinger K, Girard B, Slobod K, McPhee R, Pajon R, Aunins A, Das R, Miller JM, Schnyder Ghamloush S; KidCOVE Study Group. Evaluation of mRNA-1273 Vaccine in Children 6 Months to 5 Years of Age. N Engl J Med. 2022 Nov 3;387(18):1673-1687. doi: 10.1056/NEJMoa2209367. Epub 2022 Oct 19. PMID 36260859
- [Derived] Creech CB, Anderson E, Berthaud V, Yildirim I, Atz AM, Melendez Baez I, Finkelstein D, Pickrell P, Kirstein J, Yut C, Blair R, Clifford RA, Dunn M, Campbell JD, Montefiori DC, Tomassini JE, Zhao X, Deng W, Zhou H, Ramirez Schrempp D, Hautzinger K, Girard B, Slobod K, McPhee R, Pajon R, Das R, Miller JM, Schnyder Ghamloush S; KidCOVE Study Group. Evaluation of mRNA-1273 Covid-19 Vaccine in Children 6 to 11 Years of Age. N Engl J Med. 2022 May 26;386(21):2011-2023. doi: 10.1056/NEJMoa2203315. Epub 2022 May 11. PMID 35544369
- [Derived] Lynch LR, Clifford H, Ko R, Hache M, Sun W. Primer of COVID-19 Vaccines for the Perioperative Physician. J Neurosurg Anesthesiol. 2022 Jan 1;34(1):101-106. doi: 10.1097/ANA.0000000000000802. PMID 34870630
- See also: Click here to access the website, http://www.kidcovestudy.com, for additional information for the study, such as Study Overview, Participation, Site Locations, along with contact numbers for each location for the study. — http://www.kidcovestudy.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 3 parts: Part 1 (open-label; dose-escalation and age de-escalation), Part 2 (placebo-controlled), and Part 3 (open-label; lower dose regimen).
Pre-assignment Details: A comparison to the mRNA-1273-P301 (NCT04470427) study's efficacy data was performed on a sub-group of mRNA-1273-P301 (P301) study participants aged 18-25 (N=296). Study "Completion" and "Not Completion" data reported in the Participant Flow were collected by "Overall Study" (that is, as 1 period regardless if a booster dose was received).
Groups:
- Part 1 (6-11 Years): mRNA-1273 50 µg: Participants received 2 doses of 50 micrograms (µg) mRNA-1273 by intramuscular (IM) injection approximately 28 days apart (Day 1 and Day 29).
- Part 1 (6-11 Years): mRNA-1273 100 µg: Participants received 2 doses of 100 µg mRNA-1273 by IM injection approximately 28 days apart (Day 1 and Day 29).
- Part 1 (2-5 Years): mRNA-1273 25 µg; Part 1 (6-23 Months): mRNA-1273 25 µg; Part 2 (2-5 Years): mRNA-1273 25 µg; Part 2 (6-23 Months): mRNA-1273 25 µg: Participants received 2 doses of 25 µg mRNA-1273 by IM injection approximately 28 days apart (Day 1 and Day 29).
- Part 1 (2-5 Years): mRNA-1273 50 µg; Part 2 (6-11 Years): mRNA-1273 50 µg: Participants received 2 doses of 50 µg mRNA-1273 by IM injection approximately 28 days apart (Day 1 and Day 29).
- Part 2 (6-11 Years): Placebo: Participants received 2 doses of matching placebo by IM injection approximately 28 days apart (Day 1 and Day 29). Participants were offered crossover vaccination with 50 μg of mRNA-1273 after the availability of a coronavirus disease 2019 (COVID-19) vaccine under Emergency Use Authorization (EUA).
- Part 2 (2-5 Years): Placebo; Part 2 (6-23 Months): Placebo: Participants received 2 doses of matching placebo by IM injection approximately 28 days apart (Day 1 and Day 29). Participants were offered crossover vaccination with 25 μg of mRNA-1273 after the availability of a COVID-19 vaccine under EUA.
- Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg: Participants received 2 doses of 25 µg mRNA-1273 by IM injection approximately 28 days apart (Day 1, and Day 29).
Period: Overall Study
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg
Started | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90
Received First Injection | 380 | 371 | 75 | 149 | 150 | 997 | 3005 | 1007 | 3031 | 667 | 1993 | 90
Received Second Injection | 379 | 371 | 75 | 149 | 150 | 974 | 2995 | 984 | 3007 | 649 | 1979 | 84
Received First Injection in Open-label | 0 | 0 | 0 | 0 | 0 | 702 | 0 | 640 | 0 | 444 | 0 | 0
Received Booster Dose | 230 | 249 | 40 | 99 | 125 | 469 | 2002 | 282 | 1301 | 237 | 1016 | 70
Received Crossover Vaccination | 0 | 0 | 0 | 0 | 0 | 702 | 0 | 640 | 0 | 444 | 0 | 0
Completed | 307 | 316 | 55 | 131 | 105 | 556 | 2329 | 515 | 2086 | 366 | 1387 | 51
Not Completed | 73 | 55 | 20 | 18 | 45 | 448 | 682 | 493 | 954 | 303 | 608 | 39
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Not completed — Lost to Follow-up | 24 | 15 | 6 | 4 | 21 | 55 | 237 | 52 | 221 | 43 | 142 | 18
Not completed — Received Emergency Use Authorization (EUA) Vaccine | 5 | 4 | 0 | 3 | 1 | 194 | 37 | 222 | 29 | 115 | 9 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 3 | 18 | 1 | 7 | 0 | 5 | 0
Not completed — Withdrawal by Subject | 36 | 31 | 11 | 8 | 16 | 162 | 299 | 149 | 303 | 94 | 192 | 16
Not completed — Other Than Specified | 6 | 5 | 3 | 2 | 6 | 31 | 86 | 66 | 388 | 48 | 258 | 4
Not completed — Protocol Deviation | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 0 | 0
Not completed — Missing | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set of Part 1 and Part 3 included all dosed participants and of Part 2 included all randomized participants who received any study injection.
  Study mRNA-1273-P301 (P301) (NCT04470427) mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria.
Groups:
- Part 1 (6-11 Years): mRNA-1273 50 µg; Part 1 (2-5 Years): mRNA-1273 50 µg; Part 2 (6-11 Years): mRNA-1273 50 µg: Participants received 2 doses of 50 µg mRNA-1273 by IM injection approximately 28 days apart (Day 1 and Day 29).
- Part 2 (6-11 Years): Placebo: Participants received 2 doses of matching placebo by IM injection approximately 28 days apart (Day 1 and Day 29). Participants were offered crossover vaccination with 50 μg of mRNA-1273 after the availability of a coronavirus disease 2019 (COVID-19) vaccine under EUA.
- Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg: Participants (young adults; 18-25 years of age) received 100 μg mRNA-1273 on a 2 injection schedule in Study mRNA-1273-P301 (P301).
- Total: Total of all reporting groups
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg | Total
Number analyzed (Participants) | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90 | 296 | 12238
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P204: number analyzed (Participants) | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90 | 0 | 11942
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P204: Infants and toddlers (28 days - 23 months) | 0 | 0 | 0 | 0 | 150 | 0 | 0 | 11 | 18 | 669 | 1989 | 0 | 0 | 2837
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P204: Children (2 - 11 years) | 380 | 371 | 75 | 149 | 0 | 1004 | 3011 | 997 | 3022 | 0 | 6 | 90 | 0 | 9105
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P204: Adults (between 18 and 64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: Infants and toddlers (28 days - 23 months) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: Children (2 - 11 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Age Categorical Data for Participants Enrolled in Study mRNA-1273-P301: Adults (between 18 and 64 years) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 296
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Sex Data for Participants Enrolled in Study mRNA-1273-P204: number analyzed (Participants) | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90 | 0 | 11942
    Sex Data for Participants Enrolled in Study mRNA-1273-P204: Female | 185 | 199 | 39 | 69 | 67 | 516 | 1456 | 498 | 1490 | 341 | 981 | 34 | 0 | 5875
    Sex Data for Participants Enrolled in Study mRNA-1273-P204: Male | 195 | 172 | 36 | 80 | 83 | 488 | 1555 | 510 | 1550 | 328 | 1014 | 56 | 0 | 6067
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 153 | 153
    Sex Data for Participants Enrolled in Study mRNA-1273-P301: Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 143 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P204: number analyzed (Participants) | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90 | 0 | 11942
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P204: Hispanic or Latino | 72 | 69 | 24 | 17 | 15 | 183 | 562 | 142 | 429 | 94 | 257 | 29 | 0 | 1893
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P204: Not Hispanic or Latino | 304 | 296 | 51 | 129 | 133 | 811 | 2421 | 857 | 2593 | 568 | 1719 | 58 | 0 | 9940
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P204: Unknown or Not Reported | 4 | 6 | 0 | 3 | 2 | 10 | 28 | 9 | 18 | 7 | 19 | 3 | 0 | 109
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 78 | 78
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 216 | 216
    Ethnicity Data for Participants Enrolled in Study mRNA-1273-P301: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristics data of participants enrolled in Study mRNA-1273-P301 have been reported separately.
  Participants
    Race Data for Participants Enrolled in Study mRNA-1273-P204: number analyzed (Participants) | 380 | 371 | 75 | 149 | 150 | 1004 | 3011 | 1008 | 3040 | 669 | 1995 | 90 | 0 | 11942
    Race Data for Participants Enrolled in Study mRNA-1273-P204: White | 266 | 284 | 54 | 128 | 124 | 676 | 1960 | 793 | 2307 | 527 | 1568 | 48 | 0 | 8735
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Black or African American | 34 | 13 | 3 | 7 | 3 | 94 | 310 | 38 | 142 | 18 | 62 | 37 | 0 | 761
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Asian | 28 | 25 | 8 | 3 | 7 | 100 | 297 | 51 | 191 | 38 | 94 | 2 | 0 | 844
    Race Data for Participants Enrolled in Study mRNA-1273-P204: American Indian or Alaska Native | 0 | 2 | 0 | 0 | 1 | 3 | 15 | 3 | 11 | 0 | 7 | 2 | 0 | 44
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 5 | 0 | 0 | 0 | 0 | 13
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Other | 3 | 10 | 7 | 1 | 3 | 22 | 62 | 16 | 43 | 7 | 33 | 0 | 0 | 207
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Multiple | 39 | 31 | 3 | 10 | 11 | 98 | 330 | 100 | 324 | 76 | 215 | 0 | 0 | 1237
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Not Reported | 9 | 4 | 0 | 0 | 0 | 10 | 23 | 4 | 13 | 2 | 11 | 1 | 0 | 77
    Race Data for Participants Enrolled in Study mRNA-1273-P204: Unknown | 0 | 2 | 0 | 0 | 1 | 1 | 10 | 0 | 4 | 1 | 5 | 0 | 0 | 24
    Race Data for Participants Enrolled in Study mRNA-1273-P301: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 296 | 296
    Race Data for Participants Enrolled in Study mRNA-1273-P301: White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 207 | 207
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 29
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 30 | 30
    Race Data for Participants Enrolled in Study mRNA-1273-P301: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 14
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
    Race Data for Participants Enrolled in Study mRNA-1273-P301: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Parts 1, 2, and 3: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs)
Description: Solicited ARs were collected in an electronic diary (eDiary). Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered adverse events (AEs). Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set: all participants in Safety Set (Safety Set of Part 1 and Part 3 included all dosed participants and of Part 2 included all randomized participants who received any study injection) who contributed any solicited AR data, that is, had at least 1 post-baseline solicited safety assessment. Per prespecified analysis, data for this endpoint was not collected for the mRNA-1273.214 treatment groups.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg: Participants received a single dose of 25 μg mRNA-1273 by IM injection on Booster Dose (BD)-Day 1.
- Part 1 (6-11 Years): PS mRNA-1273 100 μg - BD 25 μg; Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 25 μg; Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 25 μg; Part 2 (6 Months-5 Yrs): PS PBO - mRNA-1273 25 μg - BD 25 μg; Part 2 (6 Months-5 Years): PS mRNA-1273 25 μg - BD 25 μg; Part 2(6-11 Yrs): PS Placebo - mRNA-1273 50 μg - BD 1273 25 μg; Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg: Participants received a single dose of 25 μg mRNA-1273 by IM injection on BD-Day 1.
- Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg; Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg; Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 10 μg: Participants received a single dose of 10 μg mRNA-1273 by IM injection on BD-Day 1.
- Part 3 (6-11 Years): BD mRNA-1273 25 µg: Participants received a third dose of 25 µg mRNA-1273 by IM injection on Day 149.
- Part 2 (6-11 Years): Placebo: Participants received 2 doses of matching placebo by IM injection approximately 28 days apart (Day 1 and Day 29). Participants were offered crossover vaccination with 50 μg of mRNA-1273 after the availability of a COVID-19 vaccine under EUA.
- Part 3 (6-11 Years): mRNA-1273 25 µg: Participants received 3 doses of 25 µg mRNA-1273 by IM injection on Days 1, 29, and 149.
Arm/Group | Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 1 (6-11 Years): PS mRNA-1273 100 μg - BD 25 μg | Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 2 (6 Months-5 Yrs): PS PBO - mRNA-1273 25 μg - BD 25 μg | Part 2 (6 Months-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 2(6-11 Yrs): PS Placebo - mRNA-1273 50 μg - BD 1273 25 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg | Part 3 (6-11 Years): BD mRNA-1273 25 µg | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): mRNA-1273 25 µg
Number analyzed (Participants) | 228 | 247 | 122 | 31 | 58 | 8 | 38 | 5 | 18 | 405 | 1853 | 56 | 380 | 371 | 69 | 153 | 150 | 994 | 3005 | 998 | 3014 | 664 | 1991 | 90
Participants | 216 | 221 | 93 | 24 | 46 | 7 | 36 | 4 | 12 | 358 | 1726 | 30 | 374 | 367 | 62 | 147 | 141 | 823 | 2983 | 797 | 2800 | 596 | 1889 | 66

2. Primary Outcome: Parts 1, 2, and 3: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. COVID-19/SARS-CoV-2 infections were considered clinical events for efficacy and not AEs. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section and presented by each dose group separately.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set of Part 1 and Part 3 included all dosed participants and of Part 2 included all randomized participants who received any study injection. Per prespecified analysis, data for this endpoint was not collected for the mRNA-1273.214 and placebo only treatment groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 1 (6-11 Years): PS mRNA-1273 100 μg - BD 25 μg | Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 2 (6 Months-5 Yrs): PS PBO - mRNA-1273 25 μg - BD 25 μg | Part 2 (6 Months-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 2(6-11 Yrs): PS Placebo - mRNA-1273 50 μg - BD 1273 25 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): mRNA-1273 25 µg
Number analyzed (Participants) | 229 | 247 | 122 | 31 | 59 | 9 | 38 | 5 | 37 | 411 | 1879 | 380 | 371 | 69 | 155 | 150 | 3007 | 3031 | 1994 | 90
Participants | 38 | 20 | 24 | 8 | 4 | 1 | 8 | 1 | 5 | 33 | 196 | 106 | 92 | 15 | 51 | 75 | 785 | 1087 | 883 | 17

3. Primary Outcome: Parts 1, 2, and 3: Number of Participants With Serious Adverse Events (SAEs), AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Discontinuation From Study
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly/birth defect, or was an important medical event. AESIs for mRNA-1273 were identified based upon medical concepts that may be related to COVID-19 or were of interest in COVID-19 vaccine safety surveillance. An MAAE is an AE that led to an unscheduled visit to a healthcare practitioner. This included visits to a study site for unscheduled assessments and visits to healthcare practitioners external to the study site. COVID-19/SARS-CoV-2 infections were considered clinical events for efficacy and not AEs. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section and presented by each dose group separately.
Time Frame: Up to 2 years
Population: Safety Set of Part 1 and Part 3 included all dosed participants and of Part 2 included all randomized participants who received any study injection. Per prespecified analysis, the data for this outcome measure was not collected for participants who received only placebo.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2(6 M-5 Yr): PS PBO - mRNA-1273 25 μg - BD 1273.214 10 μg; Part 2(6 Months-5 Yrs): PS mRNA-1273 25 μg - BD 1273.214 10 μg: Participants received a single dose of 10 μg mRNA-1273.214 by IM injection on BD-Day 1.
- Part 2(6 M-5 Yr): PS PBO - mRNA-1273 25 μg - BD 1273.214 25 μg; Part 2(6 Months-5 Yrs): PS mRNA-1273 25 μg - BD 1273.214 25 μg; Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg - BD 1273.214 25 μg; Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273.214 25 μg: Participants received a single dose of 25 μg mRNA-1273.214 by IM injection on BD-Day 1.
- Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover): Participants received a placebo in the blinded phase and then crossover vaccination with 50 μg of mRNA-1273 after the availability of a COVID-19 vaccine under EUA.
- Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover); Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover): Participants received a placebo in the blinded phase and then crossover vaccination with 25 μg of mRNA-1273 after the availability of a COVID-19 vaccine under EUA. Adverse Events were collected from the first cross-over dose until the first booster dose.
Arm/Group | Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 1 (6-11 Years): PS mRNA-1273 100 μg - BD 25 μg | Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 1 (2-5 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 2 (6 Months-5 Yrs): PS PBO - mRNA-1273 25 μg - BD 25 μg | Part 2 (6 Months-5 Years): PS mRNA-1273 25 μg - BD 25 μg | Part 2(6 M-5 Yr): PS PBO - mRNA-1273 25 μg - BD 1273.214 10 μg | Part 2(6 Months-5 Yrs): PS mRNA-1273 25 μg - BD 1273.214 10 μg | Part 2(6 M-5 Yr): PS PBO - mRNA-1273 25 μg - BD 1273.214 25 μg | Part 2(6 Months-5 Yrs): PS mRNA-1273 25 μg - BD 1273.214 25 μg | Part 2(6-11 Yrs): PS Placebo - mRNA-1273 50 μg - BD 1273 25 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg - BD 1273.214 25 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273.214 25 μg | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): mRNA-1273 25 µg | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover) | Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover) | Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover)
Number analyzed (Participants) | 229 | 247 | 122 | 31 | 59 | 9 | 38 | 5 | 37 | 505 | 2261 | 8 | 20 | 411 | 1879 | 58 | 123 | 380 | 371 | 69 | 155 | 150 | 3007 | 3031 | 1994 | 90 | 701 | 640 | 444
Participants
  SAEs | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 7 | 16 | 0 | 0 | 3 | 7 | 0 | 0 | 5 | 3 | 0 | 0 | 3 | 22 | 32 | 45 | 1 | 3 | 8 | 4
  AESIs | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 9 | 0 | 0 | 5 | 7 | 0 | 1 | 2 | 19 | 13 | 13 | 0 | 3 | 1 | 1
  MAAEs | 85 | 71 | 59 | 16 | 23 | 4 | 17 | 3 | 10 | 182 | 901 | 1 | 3 | 137 | 616 | 16 | 34 | 175 | 169 | 32 | 80 | 105 | 1095 | 1687 | 1237 | 22 | 221 | 204 | 171
  AEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Parts 1 and 2: Geometric Mean (GM) Value of Serum Pseudovirus Neutralizing Antibody ID50 Titers From Study mRNA-1273-P204 (P204) Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years) Vaccine Recipients (Day 57) in Study P301
Description: Antibody values reported as below lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ and values greater than upper limit of quantification (ULOQ) were replaced by ULOQ if actual values were not available. LLOQ was 18.5 arbitrary units (AU)/milliliter (mL) and ULOQ was 45118 AU/mL for ID50 titer. Per-Protocol (PP) Immunogenicity Subset: all enrolled participants who received planned doses of the study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment for analysis endpoint, complied with immunogenicity window based on 2nd injection timing; had negative reverse transcriptase polymerase chain reaction (RT-PCR) test for SARS-CoV-2 and negative serology test based on binding antibody (bAb) specific to SARS-CoV-2 nucleocapsid protein at baseline, not receiving highly active antiretroviral therapy (HAART) for participants with HIV; and had no major protocol deviations that impacted key or critical data.
Time Frame: Day 57 P204/Day 57 P301
Population: PP immunogenicity subset. Study P301 mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria. 'Overall number of participants analyzed' = participants evaluable for this endpoint. As planned, Part 1 immunogenicity assessment did not serve as formal noninferiority hypothesis testing. It was intended to guide the dose selection only.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 2 (6-11 Years): mRNA-1273 50 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 51 | 68 | 97 | 201 | 56 | 309 | 294
titer | 1012.5 [848.2 to 1208.6] | 1845.9 [1600.5 to 2128.9] | 1782.6 [1542.0 to 2060.7] | 1669.1 [1504.5 to 1851.6] | 1890.2 [1603.8 to 2227.7] | 1618.3 [1460.0 to 1793.9] | 1321.9 [1196.5 to 1460.5]
Statistical Analysis 1: Comparison: Part 2 (6-11 Years): mRNA-1273 50 µg vs Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg; Test type: Non-Inferiority — The noninferiority of GM value (based on GLSM) was considered demonstrated if: The lower bound of the 95% confidence interval (CI) of the geometric mean ratio (GMR) was >0.667 based on the noninferiority margin of 1.5, and the GMR point estimate ≥0.8 (minimum threshold); GMR = 1.224, 95% CI 2-sided [1.061 to 1.413]

5. Primary Outcome: Parts 2 and 3: GM Concentration of Serum Pseudovirus Neutralizing Antibody VAC62 From Study P204 Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ and values >ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset: all enrolled participants who received planned doses of the study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline in Part 2, not receiving HAART in participants with HIV; and had no major protocol deviations that impacted key/critical data. Since the number of participants enrolled in Part 3 was substantially smaller than the planned sample size required for immunogenicity hypothesis testing after Dose 2 of mRNA-1273 25 μg primary series and after a 3rd dose of mRNA-1273 25 μg, the hypothesis testing was not performed.
Time Frame: Day 57 P204/Day 57 P301
Population: PP immunogenicity subset. Study P301 mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 289 | 268 | 61 | 294
AU/mL | 1394.1 [1267.7 to 1533.1] | 1759.8 [1606.7 to 1927.4] | 4368.6 [3339.6 to 5714.6] | 1400.4 [1272.7 to 1541.0]
Statistical Analysis 1: Comparison: Part 2 (2-5 Years): mRNA-1273 25 µg; Test type: Non-Inferiority — The noninferiority of GM value (based on GLSM) was considered demonstrated if the following were true: The lower bound of the 95% CI of the GMR was >0.667 based on the noninferiority margin of 1.5, and the GMR point estimate ≥0.8 (minimum threshold); GMR = 0.995, 95% CI 2-sided [0.870 to 1.139]
Statistical Analysis 2: Comparison: Part 2 (6-23 Months): mRNA-1273 25 µg; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMR = 1.257, 95% CI 2-sided [1.101 to 1.434]

6. Primary Outcome: Parts 1 and 2: Seroresponse Rate (SRR) For Serum Pseudovirus Neutralizing Antibody ID50 From Study P204 Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Percentage of participants with seroresponse for pseudovirus neutralizing antibody ID50 are reported. Seroresponse: change from below LLOQ to equal above 4*LLOQ, or at least a 4-fold rise if baseline is ≥LLOQ. LLOQ=18.5 AU/mL and ULOQ=45118 AU/mL for ID50 titer. PP Immunogenicity Subset: all enrolled participants who received planned doses of study vaccine, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 at baseline, not receiving HAART; and had no major protocol deviations that impacted key/critical data. Since the number of participants enrolled in Part 3 was substantially smaller than the planned sample size required for immunogenicity hypothesis testing after Dose 2 of mRNA-1273 25 μg primary series and after a 3rd dose of mRNA-1273 25 μg, the hypothesis testing was not performed.
Time Frame: Day 57 P204/Day 57 P301
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): mRNA-1273 50 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 201 | 56 | 50 | 68 | 96 | 307 | 294
percentage of participants | 99.5 [97.3 to 99.9] | 100 [93.6 to 100.0] | 100 [92.9 to 100] | 100 [94.7 to 100.0] | 100 [96.2 to 100.0] | 99.0 [97.2 to 99.8] | 99.3 [97.6 to 99.9]
Statistical Analysis 1: Comparison: Part 2 (6-11 Years): mRNA-1273 50 µg; Test type: Non-Inferiority — The noninferiority of the SRR was considered demonstrated if the following were true: The lower bound of the 95% CI of the SRR difference was >-10% based on the noninferiority margin of 10% and the SRR difference point estimate was ≥-5% (minimum threshold); percentage difference = -0.3, 95% CI 2-sided [-2.2 to 1.6]

7. Primary Outcome: Parts 2 and 3: SRR For Serum Pseudovirus Neutralizing Antibody VAC62 From Study P204 Vaccine Recipients at Day 57 Compared With Those From Young Adult (18 to 25 Years of Age) Vaccine Recipients (Day 57) in Study P301
Description: Percentage of participants with seroresponse for Pseudovirus Neutralizing Antibody VAC62 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 10 and ULOQ AU/mL was 111433 AU/mL. PP Immunogenicity Subset: all enrolled participants who received planned doses of the study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment for analysis endpoint, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline in Part 2, not receiving HAART in participants with HIV; and had no major protocol deviations that impacted key or critical data.
Time Frame: Day 57 P204/Day 57 P301
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 284 | 264 | 61 | 294
percentage of participants | 98.9 [96.9 to 99.8] | 100 [98.6 to 100.0] | 88.5 [77.8 to 95.3] | 99.3 [97.6 to 99.9]
Statistical Analysis 1: Comparison: Part 2 (2-5 Years): mRNA-1273 25 µg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; percentage difference = -0.4, 95% CI 2-sided [-2.5 to 1.5]
Statistical Analysis 2: Comparison: Part 2 (6-23 Months): mRNA-1273 25 µg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; percentage difference = 0.7, 95% CI 2-sided [-0.8 to 2.4]

8. Primary Outcome: Parts 1 and 2: GM Concentration of Post-booster Dose Serum Pseudovirus Neutralizing Antibody VAC62 in Study P204 Compared With Post-primary Series (Post-Dose 2) in Young Adult (18 to 25 Years of Age) Vaccine Recipients in Study P301
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ and values greater than the ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset (Booster Dose Analysis): all enrolled participants who received 2 doses of planned doses of mRNA-1273 vaccination in Part 1 open-label phase or Part 2 blinded phase per schedule, received booster dose in Booster Dose Analysis, not receiving HAART in participants with HIV, had a negative SARS-CoV-2 status at baseline (pre-dose 1 of mRNA-1273), had BD-Day 29 Ab assessment for the analysis endpoint, no major protocol deviations that impacted key or critical data, and had not received off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: BD-Day 29 P204/Day 57 P301
Population: PP immunogenicity subset (Booster Dose Analysis). Study P301 mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria. 'Overall number of participants analyzed' = Pre-booster SARS-CoV-2 negative participants evaluable for this endpoint. 'Part 1 6-23 months group' and 'Part 1 2-5 years group' combined for noninferiority hypothesis testing. 'Part 1 and Part 2 groups of 6-11 years' combined for noninferiority hypothesis testing.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Groups:
- BD Phase Part 1 (6 Month-5 Yrs): PS mRNA-1273 25 μg - BD 10 μg: Participants received a single dose of 10 μg mRNA-1273 by IM injection on BD-Day 1.
- BD Part 1 and 2 (6-11 Yrs): PS mRNA-1273 50 μg - BD 1273 25 μg: Participants received a single dose of 25 μg mRNA-1273 by IM injection on BD-Day 1.
Arm/Group | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg | BD Phase Part 1 (6 Month-5 Yrs): PS mRNA-1273 25 μg - BD 10 μg | BD Part 1 and 2 (6-11 Yrs): PS mRNA-1273 50 μg - BD 1273 25 μg
Number analyzed (Participants) | 294 | 76 | 137
AU/mL | 1400.4 [1272.7 to 1541.0] | 5457.2 [4525.7 to 6580.3] | 5575.9 [5026.8 to 6184.9]
Statistical Analysis 1: Comparison: Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg vs BD Phase Part 1 (6 Month-5 Yrs): PS mRNA-1273 25 μg - BD 10 μg; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMR = 3.897, 95% CI 2-sided [3.158 to 4.808]
Statistical Analysis 2: Comparison: Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg vs BD Part 1 and 2 (6-11 Yrs): PS mRNA-1273 50 μg - BD 1273 25 μg; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; GMR = 3.982, 95% CI 2-sided [3.404 to 4.657]

9. Primary Outcome: Part 3: GM Concentration of Post-third Dose Serum Pseudovirus Neutralizing Antibody VAC62 in Study P204 Compared With Post-primary Series (Post-Dose 2) in Young Adult (18 to 25 Years) Vaccine Recipients in Study P301
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ and values greater than the ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset (Third Dose Analysis): all enrolled participants who received first 2 doses of planned doses of mRNA-1273 vaccination in Part 3 open-label phase per schedule, received third dose in Third Dose Analysis, not receiving HAART in participants with HIV, had BD-Day 29 antibody assessment for the analysis endpoint, had no major protocol deviations that impacted key or critical data, and had not received off-study COVID-19 vaccination prior to BD-Day 29 visit. Since the number of participants enrolled in Part 3 was substantially smaller than the planned sample size required for immunogenicity hypothesis testing after Dose 2 of mRNA-1273 25 μg primary series and after a 3rd dose of mRNA-1273 25 μg, the hypothesis testing was not performed.
Time Frame: Third Dose-Day 29 P204/Day 57 P301
Population: PP immunogenicity subset (Third Dose Analysis). Study P301 mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3 (6-11 Years): BD mRNA-1273 25 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 52 | 294
AU/mL | 4616.6 [3669.4 to 5808.3] | 1400.4 [1272.7 to 1541.0]

10. Primary Outcome: Parts 1 and 2: SRR for Post-booster Dose Serum Pseudovirus Neutralizing Antibody VAC62 From Baseline (Pre-Dose 1) Compared With Post-primary Series (Post-Dose 2) From Baseline (Pre-Dose 1) in Young Adult (18 to 25 Years) Vaccine Recipients in Study P301
Description: Percentage of participants with seroresponse for Pseudovirus Neutralizing Antibody VAC62 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset (Booster Dose Analysis): all enrolled participants who received 2 doses of planned doses of mRNA-1273 vaccination in Part 1 open-label phase or Part 2 blinded phase per schedule, received booster dose in Booster Dose Analysis, not receiving HAART in participants with HIV, had a negative SARS-CoV-2 status at baseline (pre-dose 1 of mRNA-1273), had BD-Day 29 Ab assessment for the analysis endpoint, no major protocol deviations that impacted key or critical data, and had not received off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: BD-Day 29 P204/Day 57 P301
Population: PP immunogenicity subset (Booster Dose Analysis). Study P301 mRNA-1273 100 μg: PPIS of randomly selected participants from study P301 aged 18-25 meeting pre-specified criteria. 'Overall number of participants analyzed' = Pre-booster SARS-CoV-2 negative participants evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg | BD Phase Part 1 (6 Month-5 Yrs): PS mRNA-1273 25 μg - BD 10 μg | BD Part 1 and 2 (6-11 Yrs): PS mRNA-1273 50 μg - BD 1273 25 μg
Number analyzed (Participants) | 294 | 72 | 129
percentage of participants | 99.3 [97.6 to 99.9] | 100 [95.0 to 100.0] | 100 [97.2 to 100.0]
Statistical Analysis 1: Comparison: Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg vs BD Phase Part 1 (6 Month-5 Yrs): PS mRNA-1273 25 μg - BD 10 μg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; percentage difference = 0.7, 95% CI 2-sided [-4.4 to 2.4]
Statistical Analysis 2: Comparison: Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg vs BD Part 1 and 2 (6-11 Yrs): PS mRNA-1273 50 μg - BD 1273 25 μg; Test type: Non-Inferiority — [test comment as in outcome 6, analysis 1]; percentage difference = 0.7, 95% CI 2-sided [-2.2 to 2.4]

11. Primary Outcome: Part 3: SRR for Post-third Dose Serum Pseudovirus Neutralizing Antibody VAC62 From Baseline (Pre-Dose 1) Compared With Post-primary Series (Post-Dose 2) From Baseline (Pre-Dose 1) in Young Adult (18 to 25 Years) Vaccine Recipients in Study P301
Description: Percentage of participants with seroresponse for Pseudovirus Neutralizing Antibody VAC62 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset (Third Dose Analysis): all enrolled participants who received first 2 doses of planned doses of mRNA-1273 vaccination in Part 3 open-label phase per schedule, received third dose in Third Dose Analysis, not receiving HAART in participants with HIV were not receiving HAART, had BD-Day 29 antibody assessment for the analysis endpoint, had no major protocol deviations that impacted key or critical data, and had not received off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: Third Dose-Day 29 P204/Day 57 P301
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 3 (6-11 Years): BD mRNA-1273 25 µg | Study mRNA-1273-P301 (NCT04470427) mRNA-1273 100 μg
Number analyzed (Participants) | 50 | 294
percentage of participants | 90.0 [78.2 to 96.7] | 99.3 [97.6 to 99.9]

12. Secondary Outcome: Parts 1 and 2: GM Level of Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) S Protein-specific Binding Antibody (bAb), as Measured by MesoScale Discovery (MSD) Electrochemiluminescence (ECL) Multiplex Assay on Days 1 and 57
Description: GM level of SARSCOV2S2P immunoglobulin G (IgG) antibody VAC123/VAC72, as measured by ECL multiplex assay specific to SARS-CoV-2 spike protein is reported. Antibody values reported as <LLOQ were replaced by 0.5*LLOQ and values >ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 23 AU/mL and ULOQ was 14000000 AU/mL for VAC72. LLOQ was 69 AU/mL and ULOQ was 14400000 AU/mL for VAC123. PP Immunogenicity Subset: all enrolled participants who received planned doses of study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 protein at baseline, not receiving HAART in participants with HIV; and had no major protocol deviations.
Time Frame: Day 1, Day 57 (1 month after Dose 2)
Population: PP immunogenicity subset. Overall number of participants analyzed= participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg
Number analyzed (Participants) | 200 | 56 | 50 | 68 | 96 | 308 | 304 | 285
AU/mL
  Baseline (Day 1): number analyzed (Participants) | 200 | 56 | 50 | 68 | 96 | 294 | 304 | 285
  Baseline (Day 1) | 35.6 [31.0 to 40.8] | 49.1 [33.9 to 71.1] | 15.8 [13.5 to 18.5] | 33.7 [26.2 to 43.4] | 14.6 [12.8 to 16.7] | 32.6 [28.5 to 37.3] | 24.5 [21.7 to 27.5] | 22.0 [19.1 to 25.3]
  Day 57: number analyzed (Participants) | 200 | 56 | 50 | 61 | 95 | 308 | 301 | 280
  Day 57 | 325784.0 [302917.7 to 350376.4] | 457349.2 [402424.0 to 519770.8] | 261952.0 [227935.8 to 301044.7] | 417419.8 [359399.2 to 484807.0] | 297561.7 [234740.9 to 377194.3] | 293118.9 [261748.3 to 328249.4] | 235059.2 [198610.2 to 278197.3] | 293955.4 [256077.7 to 337435.8]

13. Secondary Outcome: Parts 1 and 2: GM Level of SARS-CoV-2 S Protein-specific bAb, as Measured by MSD ECL Multiplex Assay on Baseline (Pre-dose 1), Day 57, Day 209, BD-Day 1, and BD-Day 29
Description: GM level of SARSCOV2S2P IgG antibody VAC123/VAC72 is reported. Antibody values reported as <LLOQ were replaced by 0.5*LLOQ and values >ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 23 and ULOQ was 14000000 AU/mL for VAC72. LLOQ was 69 and ULOQ was 14400000 AU/mL for VAC123. PP Immunogenicity Subset (Booster Dose Analysis): all enrolled participants who received 2 doses of planned doses of mRNA-1273 in Part 1 open-label phase or Part 2 blinded phase per schedule, received booster dose in Booster Dose Analysis, , not receiving HAART in participants with HIV, had a negative SARS-CoV-2 status at baseline, had BD-Day 29 antibody assessment for the analysis endpoint, no major protocol deviations that impacted key or critical data, and had not receive off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: Baseline (Pre-dose 1), Day 57, Day 209, BD-Day 1 (Pre-booster), BD-Day 29 (1 month after booster dose)
Population: PP immunogenicity subset (Booster Dose Analysis). Overall number of participants analyzed = participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg | Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg
Number analyzed (Participants) | 75 | 84 | 19 | 114
AU/mL
  Baseline: number analyzed (Participants) | 72 | 80 | 13 | 91
  Baseline | 50.0 [42.7 to 58.6] | 37.5 [34.3 to 40.9] | 34.5 [NA to NA] — Data not evaluable due to below limit of quantification. | 51.9 [44.6 to 60.3]
  Day 57: number analyzed (Participants) | 55 | 56 | 12 | 16
  Day 57 | 302128.3 [266991.2 to 341889.7] | 279427.6 [242953.8 to 321377.2] | 241874.9 [180565.7 to 324001.0] | 336189.6 [257789.9 to 438432.5]
  Day 209: number analyzed (Participants) | 45 | 69 | 19 | 111
  Day 209 | 74516.9 [63553.5 to 87371.5] | 66516.5 [59365.2 to 74529.2] | 71427.5 [50801.5 to 100427.9] | 85360.1 [71680.4 to 101650.5]
  BD-Day 1: number analyzed (Participants) | 75 | 77 | 19 | 114
  BD-Day 1 | 66677.7 [52382.4 to 84874.2] | 68322.4 [53860.8 to 86667.0] | 50621.5 [34112.1 to 75121.2] | 86416.4 [72836.0 to 102528.9]
  BD-Day 29: number analyzed (Participants) | 75 | 84 | 19 | 113
  BD-Day 29 | 633999.7 [561311.4 to 716101.0] | 675348.1 [584405.3 to 780443.0] | 536478.9 [403508.2 to 713268.2] | 520973.0 [469812.4 to 577704.8]

14. Secondary Outcome: Part 3: GM Level of SARS-CoV-2 S Protein-specific bAb, as Measured by MSD ECL Multiplex Assay on Baseline (Pre-dose 1), Day 57, Third Dose-Day 1, Third Dose-Day 29, Third Dose-Day 181
Description: GM level of SARSCOV2S2P IgG antibody against B.1.1.529 strain is reported. Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ and values greater than the ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 102 and ULOQ was 1180000 AU/mL for VAC123. PP Immunogenicity Subset (Third Dose Analysis): all enrolled participants who received first 2 doses of planned doses of mRNA-1273 vaccination in Part 3 open-label phase per schedule, received third dose in Third Dose Analysis, participants with HIV were not receiving HAART, had BD-Day 29 antibody assessment for the analysis endpoint, had no major protocol deviations that impact key or critical data, and had not receive off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: Baseline (Pre-dose 1), Day 57, Third Dose-Day 1, Third Dose-Day 29, Third Dose-Day 181
Population: PP immunogenicity subset (Third Dose Analysis). 'Overall number of participants analyzed = participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3 (6-11 Years): BD mRNA-1273 25 µg
Number analyzed (Participants) | 52
AU/mL
  Baseline (Pre-dose 1): number analyzed (Participants) | 50
  Baseline (Pre-dose 1) | 4659.5 [2918.7 to 7438.5]
  Day 57: number analyzed (Participants) | 50
  Day 57 | 141758.0 [118762.4 to 169206.2]
  Third Dose-Day 1: number analyzed (Participants) | 49
  Third Dose-Day 1 | 48176.2 [38955.2 to 59580.0]
  Third Dose-Day 29 | 93436.4 [77735.5 to 112308.5]
  Third Dose-Day 181: number analyzed (Participants) | 46
  Third Dose-Day 181 | 40271.7 [32950.9 to 49219.2]

15. Secondary Outcome: Parts 1 and 2: GM Value of SARS-CoV-2-specific Neutralizing Antibody ID50 Titers on Day 1 and Day 57
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ and values greater than ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. PP Immunogenicity Subset: all enrolled participants who received planned doses of the study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment for analysis endpoint, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline, not receiving HAART in participants with HIV; and had no major protocol deviations that impacted key or critical data.
Time Frame: Day 1 and Day 57 (1 month after Dose 2)
Population: PP immunogenicity subset. 'Overall number of participants analyzed' = participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): mRNA-1273 50 µg
Number analyzed (Participants) | 201 | 56 | 51 | 68 | 97 | 309
titer
  Day 1: number analyzed (Participants) | 201 | 56 | 50 | 68 | 97 | 308
  Day 1 | 9.3 [9.2 to 9.5] | 9.6 [8.9 to 10.3] | 9.3 [NA to NA] — Raw antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ in analysis. All the antibody values in these sample were below the LLOQ and were imputed identically as the value of 0.5 * LLOQ in analysis, resulting in zero variability in these samples. As a result, while geometrical mean can be calculated, the confidence intervals cannot. | 9.3 [NA to NA] — Raw antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ in analysis. All the antibody values in these sample were below the LLOQ and were imputed identically as the value of 0.5 * LLOQ in analysis, resulting in zero variability in these samples. As a result, while geometrical mean can be calculated, the confidence intervals cannot. | 9.6 [9.3 to 9.9] | 9.3 [NA to NA] — Raw antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ in analysis. All the antibody values in these sample were below the LLOQ and were imputed identically as the value of 0.5 * LLOQ in analysis, resulting in zero variability in these samples. As a result, while geometrical mean can be calculated, the confidence intervals cannot.
  Day 57 | 1669.1 [1504.5 to 1851.6] | 1890.2 [1603.8 to 2227.7] | 1012.5 [848.2 to 1208.6] | 1845.9 [1600.5 to 2128.9] | 1782.6 [1542.0 to 2060.7] | 1618.3 [1460.0 to 1793.9]

16. Secondary Outcome: Parts 2 and 3: GM Concentration of SARS-CoV-2-specific Neutralizing Antibody VAC62 on Day 1 and Day 57
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ and values greater than the ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. Data are reported per Baseline SARS-CoV-2 status: Negative and Positive. PP Immunogenicity Subset: all enrolled participants who received planned doses of the study vaccine per schedule, had baseline SARS-CoV-2 status, had baseline and Day 57 antibody assessment for analysis endpoint, complied with immunogenicity window based on 2nd injection timing; had negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline in Part 2, not receiving HAART in participants with HIV; and had no major protocol deviations that impacted key or critical data.
Time Frame: Day 1 and Day 57 (1 month after Dose 2)
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg
Number analyzed (Participants) | 315 | 311 | 57
AU/mL
  Baseline SARS-CoV-2 (Negative): Day 1: number analyzed (Participants) | 315 | 311 | 4
  Baseline SARS-CoV-2 (Negative): Day 1 | 7.9 [7.5 to 8.4] | 8.0 [7.5 to 8.5] | 21.5 [2.6 to 175.1]
  Baseline SARS-CoV-2 (Positive): Day 1: number analyzed (Participants) | 28 | 19 | 57
  Baseline SARS-CoV-2 (Positive): Day 1 | 175.3 [130.4 to 235.6] | 199.9 [109.2 to 365.9] | 177.5 [111.2 to 283.3]
  Baseline SARS-CoV-2(Negative): Day 57: number analyzed (Participants) | 298 | 278 | 4
  Baseline SARS-CoV-2(Negative): Day 57 | 1398.1 [1271.9 to 1536.8] | 1760.8 [1609.7 to 1926.0] | 2140.6 [728.7 to 6288.7]
  Baseline SARS-CoV-2 (Positive): Day 57: number analyzed (Participants) | 23 | 15 | 57
  Baseline SARS-CoV-2 (Positive): Day 57 | 7430.0 [5188.4 to 10640.1] | 10411.6 [6712.1 to 16150.1] | 4592.9 [3470.7 to 6077.9]

17. Secondary Outcome: Parts 1 and 2: GM Concentration of Post-booster SARS-CoV-2-specific Neutralizing Antibody VAC62 on Baseline, Day 57, Day 209, BD-Day 1, and BD-Day 29
Description: as for outcome 8
Time Frame: Baseline (Pre-Dose 1), Day 57 (1 month after Dose 2), Day 209 (6 months after Dose 2), BD-Day 1 (Pre-booster), and BD-Day 29 (1 month after booster dose or third dose)
Population: PP immunogenicity subset (Booster Dose Analysis). 'Overall number of participants analyzed' = participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 1 (6-23 Months): PS mRNA-1273 25 μg - BD 10 μg | Part 1 (2-5 Years): PS mRNA-1273 25 μg - BD 10 μg | Part 2 (6-11 Years): PS mRNA-1273 50 μg - BD 1273 25 μg | Part 1 (6-11 Years): PS mRNA-1273 50 μg - BD 25 μg
Number analyzed (Participants) | 84 | 19 | 114 | 75
AU/mL
  Baseline: number analyzed (Participants) | 81 | 16 | 111 | 70
  Baseline | 9.0 [8.2 to 9.9] | 12.8 [10.0 to 16.3] | 7.8 [7.1 to 8.6] | 9.3 [8.5 to 10.3]
  Day 57: number analyzed (Participants) | 56 | 18 | 18 | 55
  Day 57 | 1557.1 [1294.2 to 1873.5] | 1275.0 [983.0 to 1653.8] | 1718.7 [1316.5 to 2243.7] | 1503.3 [1292.3 to 1748.7]
  Day 209: number analyzed (Participants) | 68 | 18 | 110 | 45
  Day 209 | 448.6 [376.9 to 533.8] | 544.5 [343.1 to 864.0] | 790.7 [633.8 to 986.4] | 530.3 [432.5 to 650.2]
  BD-Day 1: number analyzed (Participants) | 75 | 18 | 113 | 75
  BD-Day 1 | 558.0 [408.5 to 762.2] | 447.2 [270.0 to 740.7] | 795.5 [640.8 to 987.5] | 627.9 [467.8 to 842.8]
  BD-Day 29 | 6474.7 [5406.0 to 7754.8] | 5778.7 [4039.7 to 8266.4] | 5805.4 [5122.4 to 6579.4] | 6991.6 [6091.2 to 8025.0]

18. Secondary Outcome: Part 3: GM Concentration of Post-third Dose SARS-CoV-2-specific Neutralizing Antibody VAC62 on Baseline, Day 57, Third Dose-Day 1, Third Dose-Day 29, and Third Dose-Day 181
Description: Antibody values reported as below the LLOQ were replaced by 0.5*LLOQ and values greater than the ULOQ were replaced by ULOQ if actual values were not available. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL. PP Immunogenicity Subset (Third Dose Analysis): all enrolled participants who received first 2 doses of planned doses of mRNA-1273 vaccination in Part 3 open-label phase per schedule, received third dose in Third Dose Analysis, not receiving HAART in participants with HIV, had BD-Day 29 antibody assessment for the analysis endpoint, had no major protocol deviations that impacted key or critical data, and had not received off-study COVID-19 vaccination prior to BD-Day 29 visit.
Time Frame: Baseline (Pre-Dose 1), Day 57 (1 month after Dose 2), Third Dose-Day 1 (at least 3 months or 6 months after Dose 2), Third Dose-Day 29 (1 month after third dose), and Third Dose-Day 181 (6 months after third dose)
Population: PP immunogenicity subset (Third Dose Analysis). 'Overall number of participants analyzed' = participants evaluable for this endpoint. Number analyzed = participants evaluable at specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part 3 (6-11 Years): BD mRNA-1273 25 µg
Number analyzed (Participants) | 52
AU/mL
  Baseline: number analyzed (Participants) | 50
  Baseline | 120.0 [71.9 to 200.3]
  Day 57: number analyzed (Participants) | 50
  Day 57 | 3775.0 [2767.5 to 5149.3]
  Third Dose-Day 1: number analyzed (Participants) | 49
  Third Dose-Day 1 | 1839.1 [1279.8 to 2643.0]
  Third Dose-Day 29 | 4616.6 [3669.4 to 5808.3]
  Third Dose-Day 181: number analyzed (Participants) | 46
  Third Dose-Day 181 | 1432.5 [1038.6 to 1975.8]

19. Secondary Outcome: Part 2: Number of Participants With SARS-CoV-2 Infection Including Symptomatic and Asymptomatic Infection (by Serology and/or RT-PCR)
Description: SARS-CoV-2 infection was defined in participants with negative SARS-CoV-2 at baseline: bAb level against SARS-CoV-2 nucleocapsid protein negative at Day 1, that became positive (as measured by Roche Elecsys) postbaseline; OR positive RT-PCR postbaseline. PP Set for Efficacy included all enrolled participants who received planned doses of study drug per schedule, complied with the 2nd injection timing, had no major protocol deviations that impacted key or critical efficacy data, and had a negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline.
Time Frame: 14 days after second injection
Population: PP set for efficacy. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg
Number analyzed (Participants) | 849 | 2606 | 854 | 2592 | 563 | 1686
Participants | 14 | 13 | 178 | 330 | 94 | 198
Statistical Analysis 1: Comparison: Part 2 (6-11 Years): Placebo vs Part 2 (6-11 Years): mRNA-1273 50 µg; Test type: Other — The 95% confidence interval (CI) of the ratio was calculated using the exact method conditional upon the total number of cases, adjusting for person-years; Vaccine Efficacy = 0.706, 95% CI 2-sided [0.325 to 0.873] — Vaccine efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 2: Comparison: Part 2 (2-5 Years): Placebo vs Part 2 (2-5 Years): mRNA-1273 25 µg; Test type: Other — The 95% CI of the ratio was calculated using the exact method conditional upon the total number of cases, adjusting for person-years; Vaccine Efficacy = 0.409, 95% CI 2-sided [0.287 to 0.509] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 3: Comparison: Part 2 (6-23 Months): Placebo vs Part 2 (6-23 Months): mRNA-1273 25 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.324, 95% CI 2-sided [0.127 to 0.474] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)

20. Secondary Outcome: Part 2: Number of Participants With Asymptomatic SARS-CoV-2 Infection, Measured by RT-PCR and/or bAb Levels Against SARS-CoV-2 Nucleocapsid Protein (by Roche Elecsys)
Description: Asymptomatic SARS-CoV-2 infection was identified by absence of symptoms and infections as detected by RT-PCR or serology tests: Absence of COVID-19 symptoms AND at least 1 from following: bAb level against SARS-CoV-2 nucleocapsid protein negative at Day 1 that became positive post-baseline, OR positive RT-PCR test post-baseline. PP Set for Efficacy included all enrolled participants who received planned doses of study drug per schedule, complied with the 2nd injection timing, had no major protocol deviations that impacted key or critical efficacy data, and had a negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline.
Time Frame: 14 days after second injection
Population: PP set for efficacy. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg
Number analyzed (Participants) | 849 | 2606 | 854 | 2592 | 563 | 1686
Participants | 10 | 10 | 55 | 124 | 21 | 70
Statistical Analysis 1: Comparison: Part 2 (6-11 Years): Placebo vs Part 2 (6-11 Years): mRNA-1273 50 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.683, 95% CI 2-sided [0.151 to 0.882] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 2: Comparison: Part 2 (2-5 Years): Placebo vs Part 2 (2-5 Years): mRNA-1273 25 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.281, 95% CI 2-sided [-0.007 to 0.480] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 3: Comparison: Part 2 (6-23 Months): Placebo vs Part 2 (6-23 Months): mRNA-1273 25 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = -0.068, 95% CI 2-sided [-0.832 to 0.352] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)

21. Secondary Outcome: Part 2: Number of Participants With Occurrence of COVID-19 (Per US Centers for Disease Control and Prevention [CDC] Case Definition of COVID-19)
Description: A COVID-19 case was identified as a positive post-baseline RT-PCR test result together with at least 1 of following systemic symptoms: fever (≥ 38 degrees Celsius [°C]/≥ 100.4 degree Fahrenheit [°F]) or chills, fatigue, headache, myalgia, nasal congestion or rhinorrhea, new loss of taste or smell, sore throat, abdominal pain, diarrhoea, nausea/vomiting, poor appetite/poor feeding; or at least 1 of following respiratory signs/symptoms: cough, shortness of breath or difficulty breathing. PP Set for Efficacy included all enrolled participants who received planned doses of study drug per schedule, complied with the 2nd injection timing, had no major protocol deviations that impacted key or critical efficacy data, and had a negative RT-PCR test for SARS-CoV-2 and negative serology test based on bAb specific to SARS-CoV-2 nucleocapsid protein at baseline.
Time Frame: 14 days after second injection
Population: PP set for efficacy.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg
Number analyzed (Participants) | 849 | 2606 | 854 | 2592 | 563 | 1686
Participants | 4 | 3 | 125 | 207 | 73 | 130
Statistical Analysis 1: Comparison: Part 2 (6-11 Years): Placebo vs Part 2 (6-11 Years): mRNA-1273 50 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.760, 95% CI 2-sided [-0.416 to 0.965] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 2: Comparison: Part 2 (2-5 Years): Placebo vs Part 2 (2-5 Years): mRNA-1273 25 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.466, 95% CI 2-sided [0.328 to 0.574] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)
Statistical Analysis 3: Comparison: Part 2 (6-23 Months): Placebo vs Part 2 (6-23 Months): mRNA-1273 25 µg; Test type: Other — [test comment as in outcome 19, analysis 2]; Vaccine Efficacy = 0.432, 95% CI 2-sided [0.232 to 0.576] — Vaccine Efficacy (percent), was defined as 1 - ratio of incidence rate (mRNA-1273 vs. placebo)

22. Other Pre Specified Outcome: Number of Deaths Related to Study Drug
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable AND/OR the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Up to 2 years
Population: Safety Set of Part 1 and Part 3 included all dosed participants and of Part 2 included all randomized participants who received any study injection. Data are reported by study part and by age categories of "6-11 years" and "6 months-5 years".
Measure: Count of Participants; unit: Participants
Groups:
- 6-11 Years: BD mRNA-1273 25 μg; 6 Months-5 Yrs: BD mRNA-1273 25 μg: Participants received a single dose of 25 μg mRNA-1273 by IM injection on BD-Day 1.
- 6-11 Yrs: BD mRNA-1273.214 25 μg; 6 Months-5 Yrs: BD mRNA-1273.214 25 μg: Participants received a single dose of 25 μg mRNA-1273.214 by IM injection on BD-Day 1.
- 6 Months-5 Yrs: BD mRNA-1273 10 μg; 6 Months-5 Yrs: BD mRNA-1273.214 10 μg: Participants received a single dose of 10 μg mRNA-1273 by IM injection on BD-Day 1.
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover) | Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover) | Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover) | Part 3 (6-11 Years): BD mRNA-1273 25 µg | 6-11 Years: BD mRNA-1273 25 μg | 6-11 Yrs: BD mRNA-1273.214 25 μg | 6 Months-5 Yrs: BD mRNA-1273 10 μg | 6 Months-5 Yrs: BD mRNA-1273 25 μg | 6 Months-5 Yrs: BD mRNA-1273.214 10 μg | 6 Months-5 Yrs: BD mRNA-1273.214 25 μg
Number analyzed (Participants) | 380 | 371 | 69 | 155 | 150 | 995 | 3007 | 1007 | 3031 | 666 | 1994 | 90 | 701 | 640 | 444 | 70 | 2766 | 184 | 212 | 89 | 2771 | 28
Participants
  Deaths | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Deaths related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Safety Set of Parts 1 & 3: dosed participants; of Part 2: randomized participants receiving study drug. Nonserious SARs persisting >7 days, leading to discontinuation or medically attended not considered AEs unless serious. COVID-19/SARS-CoV-2 infections considered clinical events for efficacy not AEs. In addition to presentation of AE data by study part, AE data are also presented by age categories "6-11 years" & "6 months-5 years" to capture AE data based on optional booster dosing.
Arm/Group | Part 1 (6-11 Years): mRNA-1273 50 µg | Part 1 (6-11 Years): mRNA-1273 100 µg | Part 1 (2-5 Years): mRNA-1273 25 µg | Part 1 (2-5 Years): mRNA-1273 50 µg | Part 1 (6-23 Months): mRNA-1273 25 µg | Part 2 (6-11 Years): Placebo | Part 2 (6-11 Years): mRNA-1273 50 µg | Part 2 (2-5 Years): Placebo | Part 2 (2-5 Years): mRNA-1273 25 µg | Part 2 (6-23 Months): Placebo | Part 2 (6-23 Months): mRNA-1273 25 µg | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover) | Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover) | Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover) | Part 3 (6-11 Years): BD mRNA-1273 25 µg | 6-11 Years: BD mRNA-1273 25 μg | 6-11 Yrs: BD mRNA-1273.214 25 μg | 6 Months-5 Yrs: BD mRNA-1273 10 μg | 6 Months-5 Yrs: BD mRNA-1273 25 μg | 6 Months-5 Yrs: BD mRNA-1273.214 10 μg | 6 Months-5 Yrs: BD mRNA-1273.214 25 μg
All-Cause Mortality (participants affected / at risk) | 0/380 | 0/371 | 0/69 | 0/155 | 0/150 | 0/995 | 0/3007 | 0/1007 | 0/3031 | 0/666 | 0/1994 | 0/90 | 0/701 | 0/640 | 0/444 | 0/70 | 0/2766 | 0/184 | 0/212 | 0/89 | 1/2771 | 0/28
Serious Adverse Events (participants affected / at risk) | 5/380 | 3/371 | 0/69 | 0/155 | 3/150 | 1/995 | 22/3007 | 3/1007 | 32/3031 | 7/666 | 45/1994 | 1/90 | 3/701 | 8/640 | 4/444 | 0/70 | 12/2766 | 0/184 | 1/212 | 1/89 | 23/2771 | 0/28
Other Adverse Events (participants affected / at risk) | 145/380 | 134/371 | 30/69 | 78/155 | 111/150 | 100/995 | 573/3007 | 356/1007 | 1341/3031 | 317/666 | 1095/1994 | 9/90 | 64/701 | 58/640 | 62/444 | 4/70 | 468/2766 | 28/184 | 56/212 | 20/89 | 655/2771 | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (6-11 Years): mRNA-1273 50 µg (N=380) | Part 1 (6-11 Years): mRNA-1273 100 µg (N=371) | Part 1 (2-5 Years): mRNA-1273 25 µg (N=69) | Part 1 (2-5 Years): mRNA-1273 50 µg (N=155) | Part 1 (6-23 Months): mRNA-1273 25 µg (N=150) | Part 2 (6-11 Years): Placebo (N=995) | Part 2 (6-11 Years): mRNA-1273 50 µg (N=3007) | Part 2 (2-5 Years): Placebo (N=1007) | Part 2 (2-5 Years): mRNA-1273 25 µg (N=3031) | Part 2 (6-23 Months): Placebo (N=666) | Part 2 (6-23 Months): mRNA-1273 25 µg (N=1994) | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg (N=90) | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover) (N=701) | Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover) (N=640) | Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover) (N=444) | Part 3 (6-11 Years): BD mRNA-1273 25 µg (N=70) | 6-11 Years: BD mRNA-1273 25 μg (N=2766) | 6-11 Yrs: BD mRNA-1273.214 25 μg (N=184) | 6 Months-5 Yrs: BD mRNA-1273 10 μg (N=212) | 6 Months-5 Yrs: BD mRNA-1273 25 μg (N=89) | 6 Months-5 Yrs: BD mRNA-1273.214 10 μg (N=2771) | 6 Months-5 Yrs: BD mRNA-1273.214 25 μg (N=28)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital hydronephrosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic disc drusen (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body ingestion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis aseptic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subperiosteal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foreign body in respiratory tract (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Greenstick fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Torus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petit mal epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disruptive mood dysregulation disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oppositional defiant disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meningitis enteroviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign rolandic epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 (6-11 Years): mRNA-1273 50 µg (N=380) | Part 1 (6-11 Years): mRNA-1273 100 µg (N=371) | Part 1 (2-5 Years): mRNA-1273 25 µg (N=69) | Part 1 (2-5 Years): mRNA-1273 50 µg (N=155) | Part 1 (6-23 Months): mRNA-1273 25 µg (N=150) | Part 2 (6-11 Years): Placebo (N=995) | Part 2 (6-11 Years): mRNA-1273 50 µg (N=3007) | Part 2 (2-5 Years): Placebo (N=1007) | Part 2 (2-5 Years): mRNA-1273 25 µg (N=3031) | Part 2 (6-23 Months): Placebo (N=666) | Part 2 (6-23 Months): mRNA-1273 25 µg (N=1994) | Part 3 (6-11 Years): Primary Series mRNA-1273 25 µg (N=90) | Part 2(6-11 Yrs): PS PBO - mRNA-1273 50 μg (Crossover) (N=701) | Part 2 (2-5 Years): PS PBO - mRNA-1273 25 μg (Crossover) (N=640) | Part 2 (6-23 Months): PBO - mRNA-1273 25 μg (Crossover) (N=444) | Part 3 (6-11 Years): BD mRNA-1273 25 µg (N=70) | 6-11 Years: BD mRNA-1273 25 μg (N=2766) | 6-11 Yrs: BD mRNA-1273.214 25 μg (N=184) | 6 Months-5 Yrs: BD mRNA-1273 10 μg (N=212) | 6 Months-5 Yrs: BD mRNA-1273 25 μg (N=89) | 6 Months-5 Yrs: BD mRNA-1273.214 10 μg (N=2771) | 6 Months-5 Yrs: BD mRNA-1273.214 25 μg (N=28)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 2 (2) | 4 (4) | 9 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Teething (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 15 (17) | 0 (0) | 1 (1) | 7 (7) | 9 (9) | 39 (43) | 109 (131) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 11 (11) | 6 (6) | 1 (1) | 6 (6) | 12 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (10) | 10 (11) | 0 (0) | 1 (1) | 9 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 17 (17) | 21 (26) | 2 (2) | 23 (29) | 40 (58) | 10 (11) | 83 (89) | 49 (58) | 222 (269) | 57 (70) | 194 (224) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 10 (10) | 2 (2) | 17 (18) | 16 (19) | 96 (107) | 15 (16) | 104 (124) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 9 (9) | 4 (4) | 3 (6) | 19 (25) | 3 (3) | 22 (22) | 47 (64) | 237 (291) | 64 (95) | 249 (353) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 37 (38) | 2 (2) | 10 (13) | 3 (4) | 141 (163) | 2 (2)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 14 (14) | 0 (0) | 8 (8) | 10 (10) | 60 (63) | 22 (22) | 114 (122) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 5 (5) | 1 (2) | 3 (3) | 7 (9) | 24 (38) | 2 (2) | 31 (35) | 42 (52) | 231 (280) | 54 (73) | 258 (385) | 0 (0) | 5 (5) | 23 (28) | 38 (45) | 0 (0) | 46 (48) | 1 (1) | 16 (22) | 5 (5) | 225 (258) | 1 (2)
Otitis media acute (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 15 (29) | 1 (1) | 12 (12) | 16 (19) | 84 (103) | 18 (24) | 113 (154) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 25 (31) | 0 (0) | 0 (0) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 8 (8) | 2 (2) | 4 (4) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 56 (87) | 50 (75) | 9 (11) | 45 (81) | 37 (70) | 47 (49) | 284 (370) | 190 (262) | 630 (926) | 146 (218) | 512 (805) | 9 (11) | 59 (64) | 39 (46) | 31 (46) | 4 (8) | 164 (205) | 2 (2) | 24 (35) | 6 (6) | 132 (142) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 11 (14) | 12 (15) | 4 (4) | 12 (13) | 9 (14) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (25) | 34 (40) | 8 (9) | 12 (14) | 27 (42) | 26 (30) | 136 (148) | 69 (90) | 262 (351) | 43 (54) | 130 (161) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 34 (45) | 5 (6) | 5 (5) | 18 (27) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 (20) | 24 (32) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 26 (31) | 6 (6) | 13 (16) | 34 (53) | 28 (30) | 107 (125) | 70 (87) | 250 (310) | 53 (70) | 173 (222) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 132 (135) | 18 (18) | 6 (7) | 3 (3) | 102 (106) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 134 (151) | 10 (12) | 12 (17) | 5 (5) | 190 (215) | 1 (2)
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 44 (44) | 1 (1) | 1 (1) | 3 (3) | 10 (10) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (3):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/96/NCT04796896/Prot_001.pdf
  • Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/96/NCT04796896/SAP_002.pdf
  • Informed Consent Form (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/96/NCT04796896/ICF_003.pdf